CLINICAL TRIAL: NCT06788938
Title: Tarlatamab in Advanced DLL3-Expressing Tumors Including Neuroendocrine Neoplasms
Brief Title: Tarlatamab in Advanced Delta-like 3 (DLL3)-Expressing Tumors Including Neuroendocrine Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-5504
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-03

CONDITIONS: DLL3-expressing Tumors; Advanced Tumors
Keywords: tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A Simon's two-stage optimum design will be used [1]. The primary objective of this phase II trial is the overall response rate (ORR, as defined by confirmed complete and partial response) per RECIST v1.1 criteria. Our null hypothesis is an ORR of 10% or lower, based on the requirements for prior therapies, and our alternative hypothesis is an ORR of 30% or greater. We will utilize a Simon two-stage design, in which 10 patients will be entered into the first stage. If 2 or more patients show a response, then an additional 19 patients will be enrolled. If 6 or more patients out of 29 show a response, then the trial will reject the null hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tarlatamab treatment (Experimental): Tarlatamab will be administered as a 60-minute intravenous (IV)
  Interventions: Drug: Tarlatamab treatment

INTERVENTIONS:
Drug: Tarlatamab treatment — * 1 mg step dose on cycle 1 day 1 (C1D1)
  * 10 mg target dose on cycle 1 day 8 (C1D8), and cycle 1 day 15 (C1D15) in a 28-day cycle.
  * 10 mg Q2W subsequently (i.e., C2 + D1/D15 dosing) in a 28-day cycle

SUMMARY:
This study is being done to learn more about the drug tarlatamab in people with your condition. The purpose of this study is to see the efficacy (how well something works) of study treatment (tarlatamab) and whether it causes any side effects. Tarlatamab is being developed as an anti-cancer drug for tumors and is FDA-approved for extensive-stage small cell lung cancer. Tarlatamab is investigational for the purpose of this study.

DETAILED DESCRIPTION:
This is a phase II, multicenter, basket trial to evaluate the safety, tolerability, and efficacy of tarlatamab in DLL3-expressing tumors. The study will enroll patients with advanced tumors, other than small cell lung cancer or neuroendocrine prostate cancer, that are confirmed to exhibit DLL3 expression. Patients will be treated with tarlatamab until disease progression, death, unacceptable adverse effects, or withdrawal of consent.

A Simon's two-stage optimum design will be used [1]. The primary objective of this phase II trial is the overall response rate (ORR, as defined by confirmed complete and partial response) per RECIST v1.1 criteria. Our null hypothesis is an ORR of 10% or lower, based on the requirements for prior therapies, and our alternative hypothesis is an ORR of 30% or greater. We will utilize a Simon two-stage design, in which 10 patients will be entered into the first stage. If 2 or more patients show a response, then an additional 19 patients will be enrolled. If 6 or more patients out of 29 show a response, then the trial will reject the null hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participant has provided informed consent prior to initiation of any study specific activities/procedures.
2. Male or female ≥ 18 years of age and willing and able to provide informed consent.
3. Histologically or cytologically confirmed malignancy other than de novo (i.e., non-transformed) SCLC or NEPC. Must be stage IV (metastatic); participants with stage III disease are eligible provided that they are not candidates for surgery and/or radiotherapy with curative intent. Acceptable tumor types include the following:

   * Low and intermediate grade neuroendocrine carcinoma (including carcinoid and atypical carcinoid)
   * Gastroenteropancreatic NEN
   * Large cell neuroendocrine carcinoma
   * SCLC transformed from previously-treated NSCLC
   * Extrapulmonary small cell carcinoma, with the exception of NEPC
   * Any other tumor type that meets staging and DLL3 positivity criteria
4. Positive DLL3 expression by immunohistochemistry on tumor biopsy.

   • Positive DLL3 expression, for purposes of this study, defined as at least 25% for participants enrolling into Stage 1 or 1% for participants enrolling into Stage 2.
5. Participants must have progressed on or following at least one line of therapy, if a standard of care therapy exists for the tumor type.
6. Measurable disease, as per RECIST 1.1
7. ECOG performance status of 0-1.
8. Adequate organ function as defined in Table 3 below. System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥ 1.0 x 109/L Platelets ≥ 100 x 109/L Hemoglobin ≥ 9 g/dL Renal Estimated glomerular filtration rate (eGFR) based on Modification of Diet in Renal Disease (MDRD) ≥ 30 mL/min/1.73 m2 Hepatic Serum total bilirubin ≤ 1.5 x ULN, with the exception of participants with Gilbert's disease AST (SGOT) and ALT (SGPT) ≤ 3 x ULN≤ 5 x ULN for patients with liver metastasis or primary liver cancer Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT), and Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy, and then only as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

Disease Related

1. Diagnosis of SCLC (with the exception of SCLC transformed from previously-treated NSCLC) or NEPC.
2. Tumor specimen is not evaluable for DLL3 expression or tumor has DLL3 surface expression < 1% by immunohistochemistry.
3. Progressive or symptomatic brain metastases. Brain metastases that have been radiated, are asymptomatic, and on a stable or decreasing dose of steroids are allowed. Leptomeningeal disease is excluded.
4. Evidence of interstitial lung disease or active, non-infectious pneumonitis. Exception: pneumonitis related to prior radiation therapy that is grade 1 and stable or improving without treatment.

   Prior/Concomitant Therapy
5. Concurrent enrollment in another clinical study, unless enrolled only in the follow-up period or an observational study. Use of any investigational anticancer therapy must not have been received within 28 days prior to the first dose of study drugs.
6. Any chemotherapy, antibody drug conjugate or immunotherapy for cancer treatment in the prior 21 days, or small molecular inhibitor in the prior 7 days.

   • Stereotactic, palliative radiation for symptomatic bone metastases is acceptable without a washout.

   • Stereotactic brain radiation for asymptomatic brain metastases is acceptable with a 7-day washout.
7. Prior therapy with any selective inhibitor of the DLL3 pathway.
8. Prior history of severe or life-threatening events from any immune-mediated therapy.
9. Receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment. Low-dose corticosteroids (prednisone ≤ 10 mg per day or equivalent is permitted)
10. Major surgical procedures within 28 days prior to first dose of study treatment.
11. Treatment with live virus, including live-attenuated vaccination, within 14 days prior to the first dose of study treatment. Inactive vaccines (e.g., non-live or non-replicating agent) and live viral non-replicating vaccines within 3 days prior to first dose of study treatment.

    Other Medical Conditions
12. History of other malignancy within the past 2 years, with the following exceptions:

    • Malignancy treated with curative intent before enrollment, with no known active disease and felt to be at low risk for recurrence by the treating physician, after discussion with the medical monitor.
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    * Adequately treated cervical carcinoma in situ without evidence of disease.
    * Adequately treated breast ductal carcinoma in situ without evidence of disease.
    * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
    * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
13. History of myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association, class II) within 6 months prior to first dose of study treatment.
14. History of arterial thrombosis (e.g., stroke or transient ischemic attack) within 6 months prior to first dose of study treatment.
15. Human immunodeficiency virus (HIV) infection.

    • Participants with HIV infection on antiviral therapy and undetectable viral load are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on study per local or institutional guidelines
16. Active hepatitis C infection.

    • Defined as participants with detectable hepatitis C antibody [HCV Ab] and hepatitis C virus [HCV] RNA viral load above the limit of quantification

    • Participants with presence of HCV antibody (HCV Ab positive) and HCV RNA viral load below the limit of quantification (HCV RNA negative) with or without prior treatment are allowed
17. Active hepatitis B infection. • Defined as presence of hepatitis B surface antigen [HBsAg-positive] and hepatitis B virus [HBV] DNA viral load above the limit of quantification [HBV DNA positive] • Participants with resolved HBV infection defined as absence of HBV surface antigen (HBsAg-negative) and presence of HBV core antibody (anti-HBc positive) followed by an HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.

    • Participants with chronic HBV infection inactive carriers state, defined as presence of HBV surface antigen (HBsAg-positive) and HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
18. Participants with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment.

    * Upon completion of antibiotics and resolution of symptoms, the participant may be considered eligible for the study from an infection standpoint.
    * Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment. Participants requiring oral antibiotics who have been afebrile > 24 hours, have no leukocytosis, nor clinical signs of infection are eligible. Screening for chronic infectious conditions is not required unless otherwise noted as exclusion criteria.

    Other Exclusions
19. Female participants of childbearing potential unwilling to use protocol specified method of contraception (see Section 5.7.2) during treatment and for an additional 60 days after the last dose of study treatment.
20. Female participants who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of study treatment.
21. Female participants planning to become pregnant or donate eggs while on study through 60 days after the last dose of study treatment.
22. Female participants of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive serum pregnancy test.
23. Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 60 days after the last dose.
24. Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of study treatment.
25. Male participants unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of study treatment.
26. Participant has known sensitivity to any of the products or components to be administered during dosing.
27. Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g., Clinical Outcome Assessments) to the best of the participant's and investigator's knowledge.
28. History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2028-04-24 (Estimated); Study Completion 2029-04-24 (Estimated)

PRIMARY OUTCOMES:
1. Primary efficacy endpoint is overall response rate (ORR) as defined as complete response (CR) or partial response (PR) by RECIST 1.1 criteria. This is evaluated in the response evaluable set of patients. | 18 months

SECONDARY OUTCOMES:
Duration of response (DOR) | 18 months
  Duration of response, defined as time from the first documentation of OR until the first documentation of disease progression or death due to any cause, whichever occurs first. Only participants who have achieved OR will be evaluated for DOR
Progression free survival (PFS) | 18 months
  Progression free survival (PFS) is defined as time from randomization until disease progression based on RECIST 1.1, or death from any cause, whichever occurs first.
Overall Survival (OS) | 18 months
  OS is defined as time from randomization until death from any cause.
Safety and tolerability | 18 months
  Safety and tolerability of tarlatamab as measured by adverse events defined by Common Terminology Criteria for Adverse Events V5.0 (CTCAE 5.0). CRS and ICANS will be graded per ASTCT Consensus Grading.

OTHER OUTCOMES:
Biomarker analysis | 18 months
  Assessment of potential biomarkers using tissue and based analyses
Evaluate radiologic correlates | 18 months
  Evaluate radiologic correlates such as DLL3 PET tracer uptake at sites where this is available.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Goldman, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (5):
- United States (5):
  - UC Davis Comprehensive Cancer Center, Davis, California
  - UCI Health Chao Family Comprehensive Cancer Center, Irvine, California
  - University of California at Los Angeles, Los Angeles, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - University of California at San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No